CLINICAL TRIAL: NCT02260193
Title: Phase 2 Open-Label Study to Assess the Efficacy, Safety, and Tolerability of AKB-6548 in Subjects With Anemia Secondary to End Stage Renal Disease (ESRD), Undergoing Chronic Hemodialysis.
Brief Title: 16-Week Repeat Oral Dose Study of AKB-6548 for Anemia in Participants With End Stage Renal Disease (ESRD) Requiring Chronic Hemodialysis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Akebia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AKB-6548-CI-0011
Record Dates: First submitted 2014-09-25; First posted 2014-10-09 (Estimated); Results first posted 2022-07-01 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Anemia; End Stage Renal Disease
Keywords: anemia; end stage renal disease; chronic kidney disease; CKD; dialysis; chronic renal insufficiency; renal impairment; erythropoietin; kidney; oral anemia treatment; hemoglobin; hypoxia-inducible factor; HIF; hypoxia-inducible factor propyl-hydroxylase inhibitor; HIF-PHI; pharmacokinetics
MeSH Terms: conditions — Anemia; Kidney Failure, Chronic; Renal Insufficiency, Chronic; Renal Insufficiency | interventions — vadadustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- AKB-6548, starting dose 1 (Experimental)
  Interventions: Drug: AKB-6548
- AKB-6548, starting dose 2 (Experimental)
  Interventions: Drug: AKB-6548
- AKB-6548, starting dose 3 (Experimental)
  Interventions: Drug: AKB-6548

INTERVENTIONS:
Drug: AKB-6548 — Starting dose 1. Oral dose administered once daily for 16 weeks. Dose adjustment based on hemoglobin level as defined in the protocol.
  Arms: AKB-6548, starting dose 1
Drug: AKB-6548 — Starting dose 2. Oral dose administered once daily for 16 weeks. Dose adjustment based on hemoglobin level as defined in the protocol.
  Arms: AKB-6548, starting dose 2
Drug: AKB-6548 — Starting dose 3. Oral dose administered three times weekly for 16 weeks. Dose adjustment based on hemoglobin levels as defined in the protocol.
  Arms: AKB-6548, starting dose 3

SUMMARY:
The purpose of this study is to evaluate the hemoglobin response (efficacy), safety, and tolerability of orally administered AKB-6548 in participants with end stage renal disease undergoing chronic hemodialysis.

ELIGIBILITY:
Key Inclusion Criteria:

* 18 to 79 years inclusive
* Chronic Kidney Disease (CKD) Stage 5 on chronic hemodialysis for at least 3 months
* Anemia secondary to CKD treated with erythropoiesis stimulating agent and intravenous iron

Key Exclusion Criteria:

* Body mass index >44.0 kilograms per meter squared (kg/m^2)
* Transfusion within 8 weeks prior to Screening
* Alanine transaminase or total bilirubin >1.25x ULN
* Uncontrolled hypertension
* Class III or IV congestive heart failure
* Myocardial infarction, acute coronary syndrome, stroke or transient ischemic attack within 6 months prior to Screening

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2014-09-10 (Actual); Primary Completion 2015-07-22 (Actual); Study Completion 2015-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Akebia Therapeutics Inc.
Locations (16):
- United States (16):
  - El Granada, California
  - Long Beach, California
  - San Dimas, California
  - Santa Clarita, California
  - Whittier, California
  - Arvada, Colorado
  - Westminster, Colorado
  - Naples, Florida
  - North Miami Beach, Florida
  - Augusta, Georgia
  - Astoria, New York
  - Arlington, Texas
  - Grand Prairie, Texas
  - Greenville, Texas
  - Houston, Texas
  - Mechanicsville, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 128 participants were screened, of which 94 participants were enrolled and randomized into the study.
Groups:
- Vadadustat 300 mg Once Daily (QD): Participants received a starting dose of Vadadustat 300 milligrams (mg) QD orally for 8 weeks. Dose increases (up to a maximum of 600 mg) were allowed once every 4 weeks after the initial 8 weeks of treatment up to Week 12, based on the changes in hemoglobin (Hgb) levels for the participant. Dose of Vadadustat were reduced at any time during the 16-week treatment period, if intolerance or an excessive increase in Hgb level (Hgb level ≥13.0 g/dL) was observed.
- Vadadustat 450 mg QD: Participants received a starting dose of Vadadustat 450 mg QD orally for 8 weeks. Dose increases (up to a maximum of 600 mg) were allowed once every 4 weeks after the initial 8 weeks of treatment up to Week 12, based on the changes in Hgb levels for the participant. Dose of Vadadustat were reduced at any time during the 16-week treatment period, if intolerance or an excessive increase in Hgb level (Hgb level ≥13.0 g/dL) was observed.
- Vadadustat 450 mg 3 Times Per Week (TIW): Participants received a starting dose of Vadadustat 450 mg TIW orally for 8 weeks. Dose increases (up to a maximum of 600 mg) were allowed once every 4 weeks after the initial 8 weeks of treatment up to Week 12, based on the changes in Hgb levels for the participant. Dose of Vadadustat were reduced at any time during the 16-week treatment period, if intolerance or an excessive increase in Hgb level (Hgb level ≥13.0 g/dL) was observed.
Period: Overall Study
Arm/Group | Vadadustat 300 mg Once Daily (QD) | Vadadustat 450 mg QD | Vadadustat 450 mg 3 Times Per Week (TIW)
Started | 30 | 33 | 31
Completed | 24 | 24 | 21
Not Completed | 6 | 9 | 10
Not completed — Lack of Efficacy | 0 | 1 | 6
Not completed — Adverse Event | 3 | 4 | 1
Not completed — Protocol Violation | 0 | 4 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 2
Not completed — Kidney Transplantation | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vadadustat 300 mg Once Daily (QD) | Vadadustat 450 mg QD | Vadadustat 450 mg 3 Times Per Week (TIW) | Total
Number analyzed (Participants) | 30 | 33 | 31 | 94
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.5 (12.44) | 59.4 (11.62) | 57.8 (8.26) | 57.6 (10.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 12 | 40
  Male | 17 | 18 | 19 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 18 | 15 | 47
  Not Hispanic or Latino | 16 | 15 | 16 | 47
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 0 | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 0 | 2
  Black or African American | 6 | 9 | 9 | 24
  White | 24 | 21 | 19 | 64
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Pre-dose Average in Hemoglobin (Hgb) Level to The Mid-study Average
Description: Change from pre-dose average was calculated by the mid-study average minus the pre-dose average. The pre-dose average was defined as the average of the 3 Hgb values that were obtained before dosing at the first screening visit, the second screening visit, and the Baseline visit; the mid-study average was defined as the average of the 2 Hgb values that were obtained at the Week 7 and Week 8 visits.
Time Frame: Pre-dose (Screening, Second Screening, and Baseline), Week 7, and Week 8
Population: Modified Intent-to-treat (MITT) Population: All participants who were assigned to study medication, received at least 1 dose of study medication, and had a pre-dose average and at least one post-baseline Hgb measurement. The primary analysis was performed in the MITT population using observed Hgb data without imputation for missing data.
Measure: Mean (Standard Deviation); unit: Grams per deciliter (g/dL)
Arm/Group | Vadadustat 300 mg Once Daily (QD) | Vadadustat 450 mg QD | Vadadustat 450 mg 3 Times Per Week (TIW)
Number analyzed (Participants) | 30 | 33 | 31
Grams per deciliter (g/dL)
  Pre-dose Average | 10.43 (0.645) | 10.55 (0.577) | 10.52 (0.534)
  Change from pre-dose average to the mid-study average: number analyzed (Participants) | 28 | 28 | 26
  Change from pre-dose average to the mid-study average | 0.00 (0.897) | -0.29 (0.970) | -0.36 (1.134)
Statistical Analysis 1: Comparison: Vadadustat 300 mg Once Daily (QD) vs Vadadustat 450 mg QD; Test type: Superiority; Least Squares Mean Differences = 0.29, 95% CI 2-sided [-0.25 to 0.82]
Statistical Analysis 2: Comparison: Vadadustat 300 mg Once Daily (QD) vs Vadadustat 450 mg 3 Times Per Week (TIW); Test type: Superiority; Least Squares Mean Differences = 0.36, 95% CI 2-sided [-0.19 to 0.90]
Statistical Analysis 3: Comparison: Vadadustat 450 mg QD vs Vadadustat 450 mg 3 Times Per Week (TIW); Test type: Superiority; Least Squares Mean Differences = 0.07, 95% CI 2-sided [-0.48 to 0.61]

2. Primary Outcome: Change From Pre-dose Average in Hgb Level to The End-of-study Average
Description: Change from pre-dose average was calculated by the end-of-study average minus the pre-dose average. The pre-dose average was defined as the average of the 3 Hgb values that were obtained before dosing at the first screening visit, the second screening visit, and the Baseline visit; the end-of-study average was defined as the average of the 2 Hgb values that were obtained at the Week 15 and Week 16 visits.
Time Frame: Pre-dose, Week 15, and Week 16
Population: MITT Population. The primary analysis was performed in the MITT population using observed Hgb data without imputation for missing data.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Vadadustat 300 mg Once Daily (QD) | Vadadustat 450 mg QD | Vadadustat 450 mg 3 Times Per Week (TIW)
Number analyzed (Participants) | 30 | 33 | 31
g/dL
  Pre-dose Average | 10.43 (0.645) | 10.55 (0.577) | 10.52 (0.534)
  Change From Pre-dose average to The End-of-study Average: number analyzed (Participants) | 24 | 24 | 21
  Change From Pre-dose average to The End-of-study Average | -0.03 (0.902) | -0.07 (0.973) | -0.14 (1.123)
Statistical Analysis 1: Comparison: Vadadustat 300 mg Once Daily (QD) vs Vadadustat 450 mg QD; Test type: Superiority; Least Squares Mean Differences = 0.04, 95% CI 2-sided [-0.54 to 0.61]
Statistical Analysis 2: Comparison: Vadadustat 300 mg Once Daily (QD) vs Vadadustat 450 mg 3 Times Per Week (TIW); Test type: Superiority; Least Squares Mean Differences = 0.10, 95% CI 2-sided [-0.49 to 0.70]
Statistical Analysis 3: Comparison: Vadadustat 450 mg QD vs Vadadustat 450 mg 3 Times Per Week (TIW); Test type: Superiority; Least squares mean difference = 0.07, 95% CI 2-sided [-0.53 to 0.66]

3. Primary Outcome: Change From Mid-study Average in Hgb Level to The End-of-study Average
Description: Change from mid-study average was calculated by the end-of-study average minus the mid-study average. The mid-study average was defined as the average of the 2 Hgb values that were obtained at the Week 7 and Week 8 visits; the end-of-study average was defined as the average of the 2 Hgb values that were obtained at the Week 15 and Week 16 visits.
Time Frame: Week 7, Week 8, Week 15, and Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Vadadustat 300 mg Once Daily (QD) | Vadadustat 450 mg QD | Vadadustat 450 mg 3 Times Per Week (TIW)
Number analyzed (Participants) | 28 | 28 | 26
g/dL
  Mid-study Average | 10.41 (0.834) | 10.26 (1.167) | 10.19 (0.950)
  Change From Mid-study Average to The End-of-study Average: number analyzed (Participants) | 24 | 24 | 21
  Change From Mid-study Average to The End-of-study Average | -0.18 (0.512) | 0.16 (0.809) | -0.07 (0.611)
Statistical Analysis 1: Comparison: Vadadustat 300 mg Once Daily (QD) vs Vadadustat 450 mg QD; Test type: Superiority; Least squares mean difference = -0.34, 95% CI 2-sided [-0.71 to 0.04]
Statistical Analysis 2: Comparison: Vadadustat 300 mg Once Daily (QD) vs Vadadustat 450 mg 3 Times Per Week (TIW); Test type: Superiority; Least squares mean difference = -0.11, 95% CI 2-sided [-0.50 to 0.29]
Statistical Analysis 3: Comparison: Vadadustat 450 mg QD vs Vadadustat 450 mg 3 Times Per Week (TIW); Test type: Superiority; Least squares mean difference = 0.23, 95% CI 2-sided [-0.16 to 0.62]

4. Secondary Outcome: Change From Baseline in Hgb
Description: Change from Baseline was calculated as the visit value minus the Baseline value. Baseline Hgb was defined as the average of the three samples obtained prior to dosing.
Time Frame: Baseline, Week 4, Week 8, Week 12, and Week 16
Population: MITT Population
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Vadadustat 300 mg Once Daily (QD) | Vadadustat 450 mg QD | Vadadustat 450 mg 3 Times Per Week (TIW)
Number analyzed (Participants) | 30 | 33 | 31
g/dL
  Baseline | 10.50 (0.702) | 10.51 (0.755) | 10.50 (0.646)
  Change from Baseline to Week 4: number analyzed (Participants) | 29 | 31 | 29
  Change from Baseline to Week 4 | -0.06 (0.708) | -0.21 (0.814) | -0.35 (0.887)
  Change from Baseline to Week 8: number analyzed (Participants) | 27 | 27 | 24
  Change from Baseline to Week 8 | -0.14 (1.058) | -0.39 (1.201) | -0.37 (1.386)
  Change from Baseline to Week 12: number analyzed (Participants) | 25 | 25 | 23
  Change from Baseline to Week 12 | 0.02 (0.995) | -0.11 (1.087) | -0.06 (1.210)
  Change from Baseline to Week 16: number analyzed (Participants) | 24 | 24 | 21
  Change from Baseline to Week 16 | -0.03 (0.946) | -0.13 (1.076) | -0.06 (1.146)

5. Secondary Outcome: Change From Baseline in Hematocrit
Description: Change from Baseline was calculated as the visit value minus the Baseline value. Baseline Hematocrit was defined as the last observation before the first dose of study medication.
Time Frame: Baseline, Week 4, Week 8, Week 12, and Week 16
Population: MITT Population
Measure: Mean (Standard Deviation); unit: Percentage of red blood cells in blood
Arm/Group | Vadadustat 300 mg Once Daily (QD) | Vadadustat 450 mg QD | Vadadustat 450 mg 3 Times Per Week (TIW)
Number analyzed (Participants) | 30 | 33 | 31
Percentage of red blood cells in blood
  Baseline | 31.2 (2.58) | 31.6 (3.75) | 31.4 (2.75)
  Change from Baseline to Week 4: number analyzed (Participants) | 29 | 31 | 29
  Change from Baseline to Week 4 | -0.4 (2.82) | -1.4 (3.36) | -0.7 (3.14)
  Change from Baseline to Week 8: number analyzed (Participants) | 27 | 27 | 24
  Change from Baseline to Week 8 | -1.0 (3.87) | -1.6 (4.73) | -1.7 (4.43)
  Change from Baseline to Week 12: number analyzed (Participants) | 25 | 25 | 23
  Change from Baseline to Week 12 | -0.2 (3.35) | -0.8 (4.07) | -0.1 (4.35)
  Change from Baseline to Week 16: number analyzed (Participants) | 24 | 24 | 20
  Change from Baseline to Week 16 | -0.8 (3.26) | -1.2 (4.19) | -0.2 (3.67)

6. Secondary Outcome: Change From Baseline in Red Blood Cell (RBC) Count
Description: Change from Baseline was calculated as the visit value minus the Baseline value. Baseline RBC Count was defined as the average of the three samples obtained prior to dosing.
Time Frame: Baseline, Week 4, Week 8, Week 12, and Week 16
Population: MITT Population
Measure: Mean (Standard Deviation); unit: 10^6 cells per microliter
Arm/Group | Vadadustat 300 mg Once Daily (QD) | Vadadustat 450 mg QD | Vadadustat 450 mg 3 Times Per Week (TIW)
Number analyzed (Participants) | 30 | 33 | 31
10^6 cells per microliter
  Baseline | 3.34 (0.278) | 3.49 (0.446) | 3.49 (0.385)
  Change from Baseline to Week 4: number analyzed (Participants) | 29 | 31 | 29
  Change from Baseline to Week 4 | -0.06 (0.235) | -0.11 (0.346) | -0.16 (0.276)
  Change from Baseline to Week 8: number analyzed (Participants) | 27 | 27 | 24
  Change from Baseline to Week 8 | -0.09 (0.357) | -0.19 (0.482) | -0.16 (0.432)
  Change from Baseline to Week 12: number analyzed (Participants) | 25 | 25 | 23
  Change from Baseline to Week 12 | -0.01 (0.325) | -0.14 (0.473) | -0.10 (0.464)
  Change from Baseline to Week 16: number analyzed (Participants) | 24 | 24 | 21
  Change from Baseline to Week 16 | -0.05 (0.309) | -0.17 (0.453) | -0.08 (0.412)

7. Secondary Outcome: Change From Baseline in Absolute Reticulocyte Count
Description: Change from Baseline was calculated as the visit value minus the Baseline value. Baseline absolute reticulocyte count was defined as the last observation before the first dose of study medication.
Time Frame: Baseline, Week 4, Week 8, Week 12, and Week 16
Population: MITT Population
Measure: Mean (Standard Deviation); unit: 10^6 cells per microliter
Arm/Group | Vadadustat 300 mg Once Daily (QD) | Vadadustat 450 mg QD | Vadadustat 450 mg 3 Times Per Week (TIW)
Number analyzed (Participants) | 30 | 33 | 31
10^6 cells per microliter
  Baseline | 0.0704 (0.02548) | 0.0661 (0.02300) | 0.0742 (0.02777)
  Change from Baseline to Week 4: number analyzed (Participants) | 28 | 31 | 29
  Change from Baseline to Week 4 | -0.0059 (0.02166) | 0.0023 (0.02597) | -0.0001 (0.02813)
  Change from Baseline to Week 8: number analyzed (Participants) | 27 | 27 | 24
  Change from Baseline to Week 8 | -0.0054 (0.01794) | 0.0041 (0.02492) | -0.0018 (0.02571)
  Change from Baseline to Week 12: number analyzed (Participants) | 21 | 25 | 23
  Change from Baseline to Week 12 | 0.0001 (0.01592) | 0.0133 (0.02734) | 0.0033 (0.02479)
  Change from Baseline to Week 16: number analyzed (Participants) | 24 | 24 | 20
  Change from Baseline to Week 16 | -0.0009 (0.02251) | 0.0048 (0.02409) | 0.0040 (0.02470)

8. Secondary Outcome: Change From Baseline in Percent Reticulocyte Count
Description: Change from Baseline was calculated as (visit value minus the Baseline value)/ Baseline value x 100. Baseline percent reticulocyte count was defined as the last observation before the first dose of study medication.
Time Frame: Baseline, Week 4, Week 8, Week 12, and Week 16
Population: MITT Population
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Vadadustat 300 mg Once Daily (QD) | Vadadustat 450 mg QD | Vadadustat 450 mg 3 Times Per Week (TIW)
Number analyzed (Participants) | 30 | 33 | 31
Percent change
  Baseline | 2.14 (0.802) | 1.89 (0.572) | 2.19 (0.927)
  Change from Baseline to Week 4 | -0.16 (0.578) | 0.14 (0.787) | 0.07 (0.884)
  Change from Baseline to Week 8 | -0.15 (0.539) | 0.24 (0.649) | 0.03 (0.710)
  Change from Baseline to Week 12 | -0.04 (0.488) | 0.48 (0.704) | 0.17 (0.835)
  Change from Baseline to Week 16 | -0.01 (0.586) | 0.23 (0.701) | 0.15 (0.817)

9. Secondary Outcome: Change From Baseline in Reticulocyte Hgb Content
Description: Change from Baseline was calculated as the visit value minus the Baseline value. Baseline reticulocyte Hgb content was defined as the average of the three samples obtained prior to dosing.
Time Frame: Baseline, Week 2, Week 4, Week 8, and Week 16
Population: MITT Population
Measure: Mean (Standard Deviation); unit: μg/dL
Arm/Group | Vadadustat 300 mg Once Daily (QD) | Vadadustat 450 mg QD | Vadadustat 450 mg 3 Times Per Week (TIW)
Number analyzed (Participants) | 30 | 33 | 31
μg/dL
  Baseline | 32.39 (1.799) | 32.12 (1.675) | 30.99 (2.372)
  Change from Baseline to Week 2: number analyzed (Participants) | 30 | 32 | 31
  Change from Baseline to Week 2 | -0.13 (1.302) | -0.03 (0.972) | 1.01 (1.621)
  Change from Baseline to Week 4: number analyzed (Participants) | 27 | 31 | 29
  Change from Baseline to Week 4 | -0.07 (0.859) | -0.21 (1.023) | 1.02 (1.425)
  Change from Baseline to Week 8: number analyzed (Participants) | 27 | 27 | 23
  Change from Baseline to Week 8 | 0.41 (1.159) | -0.27 (1.308) | 1.13 (1.301)
  Change from Baseline to Week 16: number analyzed (Participants) | 24 | 24 | 21
  Change from Baseline to Week 16 | 0.15 (1.026) | 0.58 (1.284) | -0.18 (1.494)

10. Secondary Outcome: Change From Baseline in Ferritin
Description: Change from Baseline was calculated as the visit value minus the Baseline value. Baseline ferritin was defined as the last observation before the first dose of study medication.
Time Frame: Baseline, Week 4, Week 8, Week 12, and Week 16
Population: MITT Population
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | Vadadustat 300 mg Once Daily (QD) | Vadadustat 450 mg QD | Vadadustat 450 mg 3 Times Per Week (TIW)
Number analyzed (Participants) | 30 | 33 | 31
Nanograms per milliliter (ng/mL)
  Baseline | 762.88 (470.462) | 781.96 (465.148) | 807.75 (430.981)
  Change from Baseline to Week 4: number analyzed (Participants) | 29 | 31 | 29
  Change from Baseline to Week 4 | -48.80 (205.733) | -61.21 (217.068) | -10.29 (254.574)
  Change from Baseline to Week 8: number analyzed (Participants) | 27 | 27 | 25
  Change from Baseline to Week 8 | 46.85 (529.361) | -99.11 (240.436) | -48.71 (289.063)
  Change from Baseline to Week 12: number analyzed (Participants) | 25 | 25 | 23
  Change from Baseline to Week 12 | -15.70 (316.387) | -61.81 (302.719) | 0.92 (342.188)
  Change from Baseline to Week 16: number analyzed (Participants) | 24 | 24 | 21
  Change from Baseline to Week 16 | -56.67 (317.098) | -115.36 (276.640) | -39.03 (484.937)

11. Secondary Outcome: Change From Baseline in Hepcidin
Description: Change from Baseline was calculated as the visit value minus the Baseline value. Baseline hepcidin was defined as the last observation before the first dose of study medication.
Time Frame: Baseline, Week 8, and Week 16
Population: MITT Population
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | Vadadustat 300 mg Once Daily (QD) | Vadadustat 450 mg QD | Vadadustat 450 mg 3 Times Per Week (TIW)
Number analyzed (Participants) | 30 | 33 | 31
Nanograms per milliliter (ng/mL)
  Baseline | 102.59 (58.938) | 119.61 (54.766) | 105.35 (46.805)
  Change from Baseline to Week 8: number analyzed (Participants) | 27 | 27 | 23
  Change from Baseline to Week 8 | -6.46 (49.002) | -27.80 (56.752) | -9.14 (46.498)
  Change from Baseline to Week 16: number analyzed (Participants) | 24 | 24 | 19
  Change from Baseline to Week 16 | -15.11 (46.526) | -21.66 (45.381) | -4.87 (50.379)

12. Secondary Outcome: Change From Baseline in Total Iron-Binding Capacity (TIBC)
Description: Change from Baseline was calculated as the visit value minus the Baseline value. Baseline TIBC was defined as the last observation before the first dose of study medication.
Time Frame: Baseline, Week 4, Week 8, Week 12, and Week 16
Population: MITT Population
Measure: Mean (Standard Deviation); unit: Micrograms per deciliter (μg/mL)
Arm/Group | Vadadustat 300 mg Once Daily (QD) | Vadadustat 450 mg QD | Vadadustat 450 mg 3 Times Per Week (TIW)
Number analyzed (Participants) | 30 | 33 | 31
Micrograms per deciliter (μg/mL)
  Baseline | 204.5 (39.72) | 196.7 (29.42) | 188.8 (32.28)
  Change from Baseline to Week 4: number analyzed (Participants) | 29 | 30 | 28
  Change from Baseline to Week 4 | 25.7 (21.95) | 22.0 (32.18) | 18.7 (22.39)
  Change from Baseline to Week 8: number analyzed (Participants) | 27 | 27 | 25
  Change from Baseline to Week 8 | 23.4 (28.13) | 30.3 (28.30) | 22.0 (25.37)
  Change from Baseline to Week 12: number analyzed (Participants) | 25 | 25 | 23
  Change from Baseline to Week 12 | 30.6 (30.05) | 34.8 (28.69) | 23.9 (19.62)
  Change from Baseline to Week 16: number analyzed (Participants) | 24 | 24 | 21
  Change from Baseline to Week 16 | 27.7 (35.27) | 24.9 (29.10) | 25.7 (21.78)

13. Secondary Outcome: Change From Baseline in Transferrin Saturation (TSAT)
Description: Change from Baseline was calculated as (visit value minus the Baseline value)/ Baseline value x 100. Baseline TSAT was defined as the last observation before the first dose of study medication.
Time Frame: Baseline, Week 4, Week 8, Week 12, and Week 16
Population: MITT Population
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Vadadustat 300 mg Once Daily (QD) | Vadadustat 450 mg QD | Vadadustat 450 mg 3 Times Per Week (TIW)
Number analyzed (Participants) | 30 | 33 | 30
Percent change
  Baseline | 34.6 (11.63) | 33.7 (11.14) | 37.5 (13.27)
  Change from Baseline to Week 4: number analyzed (Participants) | 29 | 29 | 28
  Change from Baseline to Week 4 | 5.4 (15.49) | 2.1 (16.97) | 3.6 (15.84)
  Change from Baseline to Week 8: number analyzed (Participants) | 27 | 27 | 24
  Change from Baseline to Week 8 | 2.9 (15.92) | 1.2 (17.31) | 3.3 (14.87)
  Change from Baseline to Week 12: number analyzed (Participants) | 25 | 25 | 23
  Change from Baseline to Week 12 | 9.1 (19.71) | 1.3 (17.18) | 3.7 (14.08)
  Change from Baseline to Week 16: number analyzed (Participants) | 24 | 24 | 21
  Change from Baseline to Week 16 | 2.5 (14.86) | 1.7 (17.44) | 2.5 (13.75)

14. Secondary Outcome: Change From Baseline in Iron
Description: Change from Baseline was calculated as the visit value minus the Baseline value. Baseline iron was defined as the last observation before the first dose of study medication.
Time Frame: Baseline, Week 4, Week 8, Week 12, and Week 16
Population: MITT Population
Measure: Mean (Standard Deviation); unit: μg/dL
Arm/Group | Vadadustat 300 mg Once Daily (QD) | Vadadustat 450 mg QD | Vadadustat 450 mg 3 Times Per Week (TIW)
Number analyzed (Participants) | 30 | 33 | 31
μg/dL
  Baseline | 70.6 (26.25) | 66.6 (23.74) | 75.4 (32.31)
  Change from Baseline to Week 4: number analyzed (Participants) | 29 | 31 | 29
  Change from Baseline to Week 4 | 20.7 (32.47) | 18.5 (40.91) | 13.3 (30.06)
  Change from Baseline to Week 8: number analyzed (Participants) | 27 | 27 | 25
  Change from Baseline to Week 8 | 14.3 (33.38) | 11.6 (39.10) | 15.0 (30.22)
  Change from Baseline to Week 12: number analyzed (Participants) | 25 | 25 | 23
  Change from Baseline to Week 12 | 31.7 (46.73) | 10.8 (31.44) | 15.5 (28.01)
  Change from Baseline to Week 16: number analyzed (Participants) | 24 | 24 | 21
  Change from Baseline to Week 16 | 14.0 (34.43) | 10.3 (37.16) | 14.0 (28.62)

15. Secondary Outcome: Number of Participants Who Received Erythropoiesis-stimulating Agent (ESA) Rescue Therapy
Description: ESA rescue therapy was administered in participants with Hgb ≤12.5 g/dL, and was stopped when Hgb reached ≥13.0 g/dL.
Time Frame: Up to Week 16
Population: Intent-to-treat (ITT) Population: All participants who were assigned to study medication and received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Vadadustat 300 mg Once Daily (QD) | Vadadustat 450 mg QD | Vadadustat 450 mg 3 Times Per Week (TIW)
Number analyzed (Participants) | 30 | 33 | 31
Participants | 4 | 6 | 2

16. Secondary Outcome: Number of Participants Who Received Blood Transfusion Rescue Therapy
Description: Blood transfusion rescue therapy was administered in participants with Hgb ≤12.5 g/dL, and was stopped when Hgb reached ≥13.0 g/dL.
Time Frame: Up to Week 16
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Vadadustat 300 mg Once Daily (QD) | Vadadustat 450 mg QD | Vadadustat 450 mg 3 Times Per Week (TIW)
Number analyzed (Participants) | 30 | 33 | 31
Participants | 1 | 1 | 0

17. Secondary Outcome: Mean Plasma Concentrations of Vadadustat
Description: Blood samples for determination of plasma levels of Vadadustat were drawn just before and 10 minutes after completion of the dialysis session.
Time Frame: Pre-dialysis and post-dialysis on Week 2 and Week 16
Population: ITT Population. Participants with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Vadadustat 300 mg Once Daily (QD) | Vadadustat 450 mg QD | Vadadustat 450 mg 3 Times Per Week (TIW)
Number analyzed (Participants) | 27 | 30 | 27
μg/mL
  Week 2 pre-dialysis | 12.89 (13.876) | 17.27 (12.741) | 5.329 (5.0281)
  Week 2 post-dialysis: number analyzed (Participants) | 26 | 30 | 27
  Week 2 post-dialysis | 13.72 (13.728) | 18.69 (15.601) | 5.287 (5.2117)
  Week 16 pre-dialysis: number analyzed (Participants) | 23 | 19 | 21
  Week 16 pre-dialysis | 11.41 (8.7716) | 15.98 (12.059) | 4.813 (3.6094)
  Week 16 post-dialysis: number analyzed (Participants) | 21 | 18 | 20
  Week 16 post-dialysis | 13.85 (11.921) | 17.38 (12.516) | 3.998 (2.9709)

18. Secondary Outcome: Mean Plasma Concentrations of Vadadustat-O-Glucuronide Metabolite
Description: as for outcome 17
Time Frame: Pre-dialysis and post-dialysis on Week 2 and Week 16
Population: ITT Population. Participants with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Vadadustat 300 mg Once Daily (QD) | Vadadustat 450 mg QD | Vadadustat 450 mg 3 Times Per Week (TIW)
Number analyzed (Participants) | 27 | 30 | 28
μg/mL
  Week 2 pre-dialysis | 16.66 (13.508) | 26.36 (21.111) | 6.295 (4.8326)
  Week 2 post-dialysis | 8.725 (7.6786) | 13.26 (13.154) | 3.101 (2.2190)
  Week 16 pre-dialysis: number analyzed (Participants) | 23 | 22 | 22
  Week 16 pre-dialysis | 15.74 (14.356) | 17.19 (13.266) | 7.843 (8.0807)
  Week 16 post-dialysis: number analyzed (Participants) | 21 | 21 | 21
  Week 16 post-dialysis | 7.833 (5.5438) | 8.408 (6.4361) | 2.998 (2.5811)

19. Secondary Outcome: Mean Plasma Concentrations of Vadadustat-Acyl-Glucuronide Metabolite
Description: as for outcome 17
Time Frame: Pre-dialysis and post-dialysis on Week 2 and Week 16
Population: ITT Population. Participants with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Vadadustat 300 mg Once Daily (QD) | Vadadustat 450 mg QD | Vadadustat 450 mg 3 Times Per Week (TIW)
Number analyzed (Participants) | 9 | 13 | 1
μg/mL
  Week 2 pre-dialysis | 0.0136 (0.00611) | 0.0224 (0.01889) | 0.0800 (NA) — Dispersion data is not available for a single participant
  Week 2 post-dialysis: number analyzed (Participants) | 9 | 10 | 0
  Week 2 post-dialysis | 0.0142 (0.01016) | 0.0095 (0.00246) |
  Week 16 pre-dialysis: number analyzed (Participants) | 9 | 3 | 0
  Week 16 pre-dialysis | 0.0129 (0.01083) | 0.0210 (0.00700) |
  Week 16 post-dialysis: number analyzed (Participants) | 6 | 3 | 0
  Week 16 post-dialysis | 0.0100 (0.00603) | 0.0087 (0.00351) |

20. Secondary Outcome: Number of Participants Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence (including a clinically significant abnormal laboratory finding) that occurred in the protocol-specified AE reporting period. A TEAE included medical conditions, signs, and symptoms not previously observed in the participant that emerged during the protocol-specified AE reporting period, including signs or symptoms associated with pre-existing underlying conditions that were not present prior to the AE reporting period. A SAE included AEs that met one or more of the following criteria/outcomes: death, lifethreatening, in-patient hospitalization or prolongation of existing hospitalization, persistent or significant disability/incapacity, and congenital anomaly/birth defect.
Time Frame: Up to Week 20
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Vadadustat 300 mg Once Daily (QD) | Vadadustat 450 mg QD | Vadadustat 450 mg 3 Times Per Week (TIW)
Number analyzed (Participants) | 30 | 33 | 31
Participants
  TEAEs | 26 | 26 | 26
  SAEs | 2 | 6 | 5

21. Secondary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Vital Signs
Description: Parameters assessed for vital signs included sitting blood pressure, pulse, respiratory rate, and body temperature. The investigator was responsible for reviewing laboratory results for clinically significant changes.
Time Frame: Up to Week 20
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Vadadustat 300 mg Once Daily (QD) | Vadadustat 450 mg QD | Vadadustat 450 mg 3 Times Per Week (TIW)
Number analyzed (Participants) | 30 | 33 | 31
Participants | 0 | 0 | 0

22. Secondary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Laboratory Parameter Values
Description: Parameters assessed for laboratory values included hematology, serum chemistry, urinalysis, iron indices, C-reactive protein, lipid profile, biomarkers, and pregnancy tests. The investigator was responsible for reviewing laboratory results for clinically significant changes.
Time Frame: Up to Week 20
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Vadadustat 300 mg Once Daily (QD) | Vadadustat 450 mg QD | Vadadustat 450 mg 3 Times Per Week (TIW)
Number analyzed (Participants) | 30 | 33 | 31
Participants | 0 | 0 | 0

23. Secondary Outcome: Number of Participants With Clinically Significant Abnormal 12-Lead Electrocardiogram (ECG) Findings
Description: A standard 12-lead ECG was performed following dosing in a supine position for approximately 5 minutes. ECGs were taken prior to vital sign assessments, circulatory access cannulation, and blood draws when possible. Clinical significance was determined by the investigator.
Time Frame: Up to Week 20
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Vadadustat 300 mg Once Daily (QD) | Vadadustat 450 mg QD | Vadadustat 450 mg 3 Times Per Week (TIW)
Number analyzed (Participants) | 30 | 33 | 31
Participants | 0 | 0 | 0

24. Other Pre Specified Outcome: Mean Intravenous Iron Replacement Therapy
Description: Intravenous iron was administered throughout the study to maintain ferritin levels in the range of ≥100 ng/mL to ≤1200 ng/mL.
Time Frame: Baseline, Week 8, and Week 16
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to Week 20 (from the time of the first dose of study medication to last dose + 4 weeks of follow-up)
Description: Treatment-emergent adverse events (TEAEs), defined as adverse events (AEs) that began (or pre-existing AEs that worsened) on or after the first dose through each participant's last participation date, were reported.
Arm/Group | Vadadustat 300 mg Once Daily (QD) | Vadadustat 450 mg QD | Vadadustat 450 mg 3 Times Per Week (TIW)
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/33 | 0/31
Serious Adverse Events (participants affected / at risk) | 5/30 | 9/33 | 8/31
Other Adverse Events (participants affected / at risk) | 22/30 | 19/33 | 23/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vadadustat 300 mg Once Daily (QD) (N=30) | Vadadustat 450 mg QD (N=33) | Vadadustat 450 mg 3 Times Per Week (TIW) (N=31)
Acute myocardial infarction (Cardiac disorders) | 1 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1 | 1
Arteriovenous fistula site infection (Infections and infestations) | 0 | 0 | 1
Abscess limb (Infections and infestations) | 0 | 1 | 0
Arteriovenous graft site infection (Infections and infestations) | 0 | 1 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0 | 0
Vestibular neuronitis (Infections and infestations) | 0 | 1 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 | 0 | 1
Delayed recovery from anaesthesia (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vadadustat 300 mg Once Daily (QD) (N=30) | Vadadustat 450 mg QD (N=33) | Vadadustat 450 mg 3 Times Per Week (TIW) (N=31)
Hyperparathyroidism secondary (Endocrine disorders) | 0 (0) | 0 (0) | 3 (3)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 4 (4) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 4 (6) | 2 (3)
Nausea (Gastrointestinal disorders) | 4 (4) | 3 (4) | 4 (5)
Vomiting (Gastrointestinal disorders) | 3 (3) | 3 (4) | 3 (3)
Fatigue (General disorders) | 2 (2) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 2 (2) | 0 (0) | 0 (0)
Pain (General disorders) | 2 (2) | 0 (0) | 1 (2)
Pyrexia (General disorders) | 1 (1) | 3 (3) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 3 (6) | 0 (0) | 0 (0)
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
Procedural hypotension (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 1 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 3 (3) | 2 (2)
Headache (Nervous system disorders) | 3 (3) | 2 (2) | 3 (4)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 2 (2) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No